CLINICAL TRIAL: NCT02520232
Title: Pathological and Non-pathological Aging, Physical Activity, Genotype and Cognition (VIAGECO)
Brief Title: Pathological and Non-pathological Aging, Physical Activity, Genotype and Cognition
Acronym: VIAGECO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Poitiers University Hospital (Other); Centre National de la Recherche Scientifique, France (Other); University of Poitiers (Other); University of Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CHUBX 2013/22
Record Dates: First submitted 2015-07-31; First posted 2015-08-11 (Estimated); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Alzheimer's Disease
Keywords: chronic exercise; genetic polymorphisms; brain imagery; executive functions; alzheimer's disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Physical activity program (A) (Experimental): Physical exercises
  Interventions: Behavioral: Combination of aerobic and strength exercises
- Physical activity program (B) (Experimental): Physical exercises
  Interventions: Behavioral: Stretching and balance exercise program
- Control (No Intervention): No physical exercices assigned by the protocol

INTERVENTIONS:
Behavioral: Combination of aerobic and strength exercises — Combination of aerobic and strength exercises
  Arms: Physical activity program (A)
Behavioral: Stretching and balance exercise program — Stretching and balance exercise program
  Arms: Physical activity program (B)

SUMMARY:
Alzheimer's disease (AD) is an irreversible, progressive brain disease. It is the most common form of dementia and the major cause of functional dependence in the elderly. Since there is currently no cure for Alzheimer's disease, a growing number of scientists pointed out the interest to use non-pharmacological alternative therapeutic approaches in order to slow down the decline of physical and cognitive resources and improve quality of life of patients with Alzheimer's disease. Several narrative and meta-analytical reviews suggest that regular practice of physical activity delays the occurrence of cognitive decline and slows down Alzheimer's disease progress when compared with sedentary people. Despite the growing interest of the scientific community for the positive effects of chronic exercise on mental health and cognitive functions, the clinical reality of this phenomenon remains to be clearly established, more particularly in aged people suffering from neurodegenerative diseases.The first aim of this research project is to test if chronic exercise reduces and even compensates for a cognitive decline in both patients with prodromal Alzheimer's disease (i.e., no dementia) and aging people with no pathology of central nervous system. The second aim of this research project is to examine whether an increasing of cerebral blood flow induced by chronic exercise can explain this positive effect.

DETAILED DESCRIPTION:
Several epidemiologic studies conducted in North America and in Europe have shown that the regular practice of physical activity, in opposition to a sedentary life, is associated with a reduced risk of developing neurodegenerative diseases such as AD. These results have been strengthened by cross-sectional and interventional studies, which have shown that physical activity slows down the decline of cognitive functions typically observed in normal and pathological aging and retards the onset of dementia. The positive effects of chronic exercise on cerebral and cognitive ageing are now recognised by scientists and clinicians; however, the mechanisms underlying these effects in humans are poorly understood and there is a real need for randomised controlled trial (RCT) on this topic. The objective of this research project is to understand the compensatory mechanisms that may account for the positive effects of regular physical activity on pathological and non-pathological cerebral ageing in human and in particular in people presenting prodromal AD. All participants will be separated into six groups corresponding to the combination of two independent variables: the population type (aged people without any neurological disease vs. prodromal Alzheimer's disease participants) and the type of physical activity program they will follow during six months (aerobic and strength exercise program, stretching and balance program, or maintaining sedentary life style). Cognitive performance, cardiovascular health, brain integrity and cerebral functioning will be assessed at two or three different times: before the onset of the training program (pre-test), at the end of the training period (post-test 1) and six months after the end of the training program (post-test 2).

ELIGIBILITY:
Inclusion Criteria:

* Aged between 60 and 80 years
* Retired
* Complete autonomy on the following four instrumental activities of daily living scales (IADL) : ability to use telephone, mode of transportation, responsibility for own medications and ability to handle finances, level of physical activity practice ≤ 2
* 18.5 ≤ BMI < 40
* MMSE ≥ 25
* For prodromal Alzheimer Disease patients : subjective memory complaints of the participant, objective evidence of impaired encoding in episodic memory (Grober-Buschke free recall score < 17).

Exclusion Criteria:

* Presence of a counter-indication for Magnetic Resonance Imaging , presence of a counter-indication for Positron Emission TomographyScan with [18F]-Flutemetamol, presence of any health problem preventing travel to the imaging service of the University Hospital, being under the legal guardianship of another person or being unable to provide consent to participate

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-02-10 (Actual); Study Completion 2018-05-11 (Actual)

PRIMARY OUTCOMES:
Executive functions (Mean z score) | 0 to 3 months after inclusion visit
  Mean z score of performances in five tasks involving executive functions (Trail Making Test, Random Number Generation Task, Stroop Color Word Test, Eriksen's Flanker Task, Letter Running Span Task).
Executive functions (Mean z score) | 6 to 9 months after inclusion visit
Executive functions (Mean z score) | 12 to 15 months after inclusion visit

SECONDARY OUTCOMES:
Senior Fitness Test score | 0 to 3 months after inclusion visit ; 6 to 9 months after inclusion visit ; 12 to 15 months after inclusion visit
Body Mass Index | Day 0 (Inclusion visit)
Energy expenditure related to physical activity (Actimetry) | 3 to 6 months after inclusion visit
  Actimetry meseare
Heart rate variability at rest | 0 to 3 months after inclusion visit ; 6 to 9 months after inclusion visit ; 12 to 15 months after inclusion visit
Blood pressure | 0 to 3 months after inclusion visit ; 6 to 9 months after inclusion visit ; 12 to 15 months after inclusion visit
Depression score | 0 to 3 months after inclusion visit ; 6 to 9 months after inclusion visit ; 12 to 15 months after inclusion visit
Self-efficacy score | 0 to 3 months after inclusion visit ; 6 to 9 months after inclusion visit ; 12 to 15 months after inclusion visit
Quality of life score | 0 to 3 months after inclusion visit ; 6 to 9 months after inclusion visit ; 12 to 15 months after inclusion visit
Stage of change score related to physical activity | 0 to 3 months after inclusion visit ; 6 to 9 months after inclusion visit ; 12 to 15 months after inclusion visit
Score at Verbal working-memory span | 0 to 3 months after inclusion visit ; 6 to 9 months after inclusion visit ; 12 to 15 months after inclusion visit
Reaction time in a two-choice reaction time task | 0 to 3 months after inclusion visit ; 6 to 9 months after inclusion visit ; 12 to 15 months after inclusion visit
Error rate in a two-choice reaction time task | 0 to 3 months after inclusion visit ; 6 to 9 months after inclusion visit ; 12 to 15 months after inclusion visit
Logic memory score | 0 to 3 months after inclusion visit ; 6 to 9 months after inclusion visit ; 12 to 15 months after inclusion visit
Grey and white matter volumes in regions of interest | 0 to 3 months after inclusion visit ; 6 to 9 months after inclusion visit
Cerebral perfusion in the same regions of interest | 0 to 3 months after inclusion visit ; 0 to 15 days after inclusion visit ; 6 to 9 months after inclusion visit
  Brain Imaging
Resting State Networks Activity | 0 to 3 months after inclusion visit ; 0 to 15 days after inclusion visit ; 6 to 9 months after inclusion visit
  Brain Imaging
Brain glucose metabolism | 0 to 3 months after inclusion visit ; 0 to 15 days after inclusion visit ; 6 to 9 months after inclusion visit
  Brain Imaging

CONTACTS AND LOCATIONS:
Overall Officials: Michèle ALLARD, Principal Investigator — University Hospital, Bordeaux; Michel AUDIFFREN, Study Chair — CNRS Poitiers; Hélène AMIEVA, Study Chair — University of Bordeaux
Locations (2):
- France (2):
  - University Hospital Bordeaux, France, Bordeaux
  - University Hospital, Poitiers, Poitiers